CLINICAL TRIAL: NCT02112422
Title: The Role of Timing of Dexamethasone Administration on Pain Scores and Quality of Recovery in Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Duane Funk, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2013:159
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Pregnancy
Keywords: Parturients
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients in the intervention group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline 45-60 minutes prior to the OR. The control group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline immediately prior to skin incision.
  Interventions: Drug: Control
- Intervention (Experimental): Patients in the intervention group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline 45-60 minutes prior to the OR. The control group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline immediately prior to skin incision.
  Interventions: Drug: Intervention

INTERVENTIONS:
Drug: Control — The control group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline immediately prior to skin incision.
  Other Names: 0.15 mg/kg dexamethasone IV prior to skin incision.
  Arms: Control
Drug: Intervention — Patients in the intervention group will receive 0.15 mg/kg of intravenous dexamethasone (maximum dose 20mg) in 100ml normal saline 45-60 minutes prior to the OR.
  Other Names: 0.15 mg/kg of dexamethasone IV 60 minutes prior to the OR.
  Arms: Intervention

SUMMARY:
The purpose of our study was to evaluate the hypothesis that single dose dexamethasone given sixty minutes preoperatively reduces visual analog scale (VAS) pain scores and improves quality of recovery in patients undergoing elective cesarean section as compared to the same dose given immediately prior to skin incision.

DETAILED DESCRIPTION:
Dexamethasone, a potent synthetic glucocorticoid with minimal mineralocorticoid effects, is commonly administered as an anesthesia adjunct for the prevention of postoperative nausea and vomiting (PONV). Over the last two decades the analgesic effects of dexamethasone have also been demonstrated in the treatment of acute and chronic pain. Two recent meta-analyses of over thirty randomized clinical trials (close to 5,000 subjects) concluded that dexamethasone at doses more than 0.1 mg/kg is an effective adjunct in multimodal strategies to reduce postoperative pain and opioid consumption after a variety of surgeries.

Cesarean section is a common surgical procedure and associated with a moderate amount of postoperative pain (Visual analogue score (VAS) of 3-5, on a 10 point scale). Patients' postoperative experience closely correlates with their perception of pain management. Controlling postoperative pain after cesarean section remains an important clinical challenge. A multimodal approach to reduce pain has become a standard of care and includes varying doses of intrathecal local anesthetic, intrathecal morphine, co-administration of opioids or other adjuncts such as non-steroidal anti-inflammatory drugs and acetaminophen. Dexamethasone is typically administered in the elective cesarean section population for the prevention of intrathecal opioid induced PONV. Recently however, the potential benefit of single dose dexamethasone has been demonstrated in improving postoperative analgesia in this patient population.

The analgesic effect of dexamethasone in post-cesarean section parturients is likely to be mediated via its anti-inflammatory actions. This does not come as a surprise given the profound inflammatory changes associated with the peripartum period and cesarean sections. Until the late third trimester. pregnancy is thought to be associated with suppression of a variety of humoral and cell-mediated immunological functions to accommodate the "foreign" semi-allogeneic fetal graft. The proinflammatory milleu becomes up regulated in late pregnancy and around the time of delivery. Specifically, during the third trimester, the percentage of granulocytes and cluster of differentiation 8 (CD8+) T lymphocytes are significantly increased, along with a concomitant reduction in the percentages of cluster of differentiation 4 (CD4+) T lymphocytes and monocytes. During the peripartum and delivery period, leukocyte count may become markedly elevated, attaining levels of 25,000/μL or greater. Moreover, circulating leukocytes undergo significant phenotypic changes including the upregulation of adhesion molecules. Other markers of inflammation including C-reactive protein, erythrocyte sedimentation rate (ESR) and complement factors C3 and C4 are all increased in normal pregnancy and significantly so during labour.

Cesarean section itself causes significant surgical stress and results in a profound inflammatory response. Inflammation is triggered not only by direct tissue injury from surgical incision and deeper tissue trauma but also by "spillage" of highly pro-inflammatory mediators from amniotic fluid and placental tissue into the pelvic cavity as well as systemic circulation.

As a result of the inflammatory insults of pregnancy and cesarean section, dexamethasone has emerged as an important adjunct in postoperative pain control in this patient population. Unanswered, however, is the role that the timing of dexamethasone administration may play in its analgesic action. Dexamethasone peak effect is delayed by 60-90 minutes reflecting its unique pharmacodynamics. Unbound dexamethasone crosses cell membranes and binds with high affinity to specific cytoplasmic glucocorticoid receptors. This complex binds to DNA elements (glucocorticoid response elements) which results in a modification of transcription and protein synthesis. This leads to inhibition of leukocyte infiltration at the site of inflammation, interference in the function of mediators of inflammatory response, suppression of humoral immune responses, and reduction in edema or scar tissue. Direct anti-inflammatory actions of dexamethasone are thought to involve phospholipase A2 inhibitory proteins and lipocortins (which control the biosynthesis prostaglandins and leukotrienes). This multistep mechanism of action may explain why administration of dexamethasone prior to the stress of surgery may optimize its therapeutic effects including analgesia and anti-emesis. However, the vast majority of studies on dexamethasone administer the drug immediately prior to or during surgery.

The purpose of this randomized, double-blinded trial is to determine if single dose dexamethasone given 45-60 minutes preoperatively reduces VAS pain scores and improves quality of recovery in patients undergoing elective cesarean section as compared to the same dose given immediately after surgical incision.

ELIGIBILITY:
Inclusion Criteria:

* •Over 18 years of age

  * American Society of Anesthesiologists class I-III
  * Presenting for elective cesarean section.

Exclusion Criteria:

* •Contraindication to regional anesthesia

  * Allergy to study drug
  * Uncontrolled diabetes
  * Active infection
  * Adrenal axis pathology
  * Active treatment with steroids
  * Treatment with oral or parenteral steroids within the previous 6 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain using visual analogue score. | 24 hours

SECONDARY OUTCOMES:
Number of episodes of Nausea and Vomiting | 24 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Duane J Funk, MD FRCP(C), Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Health Sciences Center, Winnipeg, Manitoba
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba